CLINICAL TRIAL: NCT00014118
Title: A Phase II Trial OF Chemoradiation For Organ Preservation In Resectable Stage III or IV Squamous Cell Carcinomas Of The Larynx Or Oropharynx
Brief Title: Chemotherapy and Radiation Therapy in Treating Patients With Stage III or Stage IV Larynx or Oropharynx Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068468; U10CA021115 (NIH); ECOG-2399
Record Dates: First submitted 2001-04-10; First posted 2003-01-27 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Carboplatin; Paclitaxel; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy followed by radiation therapy and chemotherapy in treating patients who have stage III or stage IV cancer of the larynx or stage III or stage IV cancer of the oropharynx.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the organ preservation rate in patients with stage III or IV squamous cell carcinoma of the larynx or oropharynx treated with paclitaxel and carboplatin followed by paclitaxel with concurrent radiotherapy.
* Determine the feasibility and toxicity of this regimen in these patients.
* Determine the utility of pre- and post-treatment organ function instruments on swallowing ability and voice quality in patients treated with this regimen.
* Determine the disease-free survival and patterns of failure of patients treated with this regimen.
* Determine the objective tumor response rate (complete and partial response) in these patients following treatment with 2 courses of induction therapy with paclitaxel and carboplatin.
* Determine changes in quality of life of patients treated with this regimen.
* Determine whether the presence of human papilloma virus infection and p-glycoprotein correlates with outcome in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to disease site (larynx vs oropharynx).

Patients receive induction therapy comprising paclitaxel IV over 3 hours followed by carboplatin IV over 30-60 minutes on days 1 and 22. Within 28 days after completion of induction therapy, patients with responding or stable disease receive paclitaxel IV over 60 minutes on days 1, 8, 15, 22, 29, 36, and 43 and radiotherapy once daily, 5 times weekly, for 7 weeks beginning on day 1.

Within 6-8 weeks after completion of therapy, patients who initially had bulky neck disease (N3) or who have residual palpable lymphadenopathy undergo surgical neck dissection. Patients with N1-N2 disease with complete response may also undergo neck dissection. Patients with initial complete response who recur at the primary site undergo surgical salvage.

Quality of life is assessed at baseline, after induction therapy, and at 3, 12, and 24 months after completion of all therapy.

Patients are followed at 6 weeks, 3 months, every 6-8 weeks for 1 year, every 3 months for 1 year, every 4 months for 1 year, and then every 6 months for 5 years thereafter.

PROJECTED ACCRUAL: A total of 110 patients (55 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage III or IV (T2-T4) squamous cell carcinoma of the larynx or oropharynx

  * No recurrent disease
  * No evidence of distant metastasis
* Resectable disease, defined as follows:

  * High probability of attaining clear surgical margins (for disease of the base of tongue, tonsil, soft palate, or pharyngeal wall)
  * No extension to root of tongue (for disease of the base of tongue)
  * No extension into pterygoid by radiograph (for disease of the tonsil, soft palate, or pharyngeal wall)
  * No primary tumor or nodal metastases fixed to the carotid artery or cervical spine (for disease of the base of tongue, tonsil, soft palate, or pharyngeal wall)
  * No trismus (for disease of the tonsil, soft palate, or pharyngeal wall)
  * No involvement of the trachea greater than 1 cm or any involvement of the esophagus (for disease of the subglottis)
  * For disease of the supraglottis, glottis, or subglottis:

    * No base of the tongue invasion greater than 2 cm
    * No tumor extension through cartilage to involve strap muscles of the neck
    * No tumor fixation to prevertebral fascia
    * No involvement of the carotid artery
    * No fixed nodal disease with involvement of the deep neck
    * Extension into pyriform sinus or lateral pharyngeal wall allowed if no extension into posterior pharynx
* Measurable disease

  * - Lesions accurately measured in at least one dimension as > 20 mm (2.0 cm) with conventional techniques or as > 10 mm (1.0 cm) with spiral CT scan
  * Cytologic or histologic evidence of neoplasm is needed for measurable disease restricted to a solitary lesion
* No other concurrent head and neck neoplasms

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Not specified

Renal

* Creatinine less than 3.0 mg/dL
* Calcium normal

Cardiovascular

* No significant cardiac disease
* No uncontrolled hypertension
* No unstable angina
* No congestive heart failure
* No myocardial infarction within the past year
* No serious cardiac arrhythmias requiring medication

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after study completion
* No significant detectable infection
* No history of allergy to drugs containing Cremophor EL
* No history of allergy to mammalian cell-derived products (epoetin alfa) or human albumin
* No other malignancy within the past 3 years except basal or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy
* No concurrent amifostine

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy above the clavicles

Surgery

* No prior surgery to the primary tumor except biopsy or debulking

Other

* No concurrent experimental mucosal protectants

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-06-06 (Actual); Primary Completion 2007-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Organ preservation rate
Feasibility and toxicity
Utility of pre- and post-treatment organ function instruments
Disease-free survival and patterns of failure
Objective tumor response rate (complete and partial response)
Changes in quality of life
Correlation of the presence of human papilloma virus infection and p-glycoprotein with outcome

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J. Cmelak, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (47):
- United States (47):
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Watson Clinic, LLC, Lakeland, Florida
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Hematology/Oncology of the North Shore at Gross Point Medical Center, Skokie, Illinois
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin

REFERENCES:
- [Result] Fakhry C, Westra WH, Li S, Cmelak A, Ridge JA, Pinto H, Forastiere A, Gillison ML. Improved survival of patients with human papillomavirus-positive head and neck squamous cell carcinoma in a prospective clinical trial. J Natl Cancer Inst. 2008 Feb 20;100(4):261-9. doi: 10.1093/jnci/djn011. Epub 2008 Feb 12. PMID 18270337
- [Result] Cmelak AJ, Li S, Goldwasser MA, Murphy B, Cannon M, Pinto H, Rosenthal DI, Gillison M, Forastiere AA. Phase II trial of chemoradiation for organ preservation in resectable stage III or IV squamous cell carcinomas of the larynx or oropharynx: results of Eastern Cooperative Oncology Group Study E2399. J Clin Oncol. 2007 Sep 1;25(25):3971-7. doi: 10.1200/JCO.2007.10.8951. PMID 17761982
- [Result] Fakhry C, Westra W, Li S, et al.: Prognostic significance of human papillomavirus (HPV) tumor status for patients with head and neck squamous cell carcinoma (HNSCC) in a prospective, multi-center phase II clinical trial. [Abstract] J Clin Oncol 25 (Suppl 18): A-6000, 299s, 2007.
- [Result] Cmelak AJ, Li S, Murphy B, et al.: Locally advanced resectable larynx (L) or oropharynx (OP) cancer: updated results of organ preservation trial ECOG 2399. [Abstract] J Clin Oncol 24 (Suppl 18): A-5527, 286s, 2006.
- [Result] Murphy BA, Smith K, Cmelak A, et al.: Swallowing function for patients treated on E2399: a phase II trial of function preservation with induction paclitaxel/carboplatin followed by radiation plus weekly paclitaxel. [Abstract] J Clin Oncol 24 (Suppl 18): A-5524, 2006.
- [Result] Murphy BA, Smith K, Dowling E, et al.: Baseline swallowing function for patients treated on E2399: a phase II trial of function preservation with induction paclitaxel/carboplatin followed by radiation plus weekly paclitaxel. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-2005, 2003.